CLINICAL TRIAL: NCT05366985
Title: Digital Evaluation of the Early Volumetric Changes of the Labial Alveolar Contour Following Guided Socket Shield Technique for Immediate Implant Placement: A Clinical Study
Brief Title: Dimensional Changes of the Labial Alveolar Ridge After Socket Shield Technique With Computer Guided Root Sectioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharos University in Alexandria (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Sameh Nabawi, Principal Investigator, Pharos University in Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07071992
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Edentulous Alveolar Ridge; Dental Trauma
Keywords: Bone implant interactions; Periodontology,; Soft tissue-implant interactions; Surgical techniques; Wound healing
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Socket shield with guided root sectioning (Experimental): Tooth extraction and immediate implant placement using the socket shield technique with computer guided sectioning of the root.
  Interventions: Procedure: Socket shield technique with computer guided sectioning of the root

INTERVENTIONS:
Procedure: Socket shield technique with computer guided sectioning of the root — A computer guide was used to section the root, leaving the coronal 2/3 of its labial part attached to the socket. An implant was then placed.
  Preoperative and Postoperative (5 months later) intraoral scans were superimposed with a digital software to assess the dimensional changes of the labial alveolar ridge. Linear changes at 1,3 and 5 mm from the gingival margin and mean linear changes in a specified Area Of Interest (AOI) were measured

SUMMARY:
In this study, the dimensional changes of the labial alveolar ridge are digitally assessed after immediate implant placement using the socket shield technique with computer guided sectioning of the root.

DETAILED DESCRIPTION:
Ten hopeless teeth in the esthetic zone were included. A computer guide was used to section the root, leaving the coronal 2/3 of its labial part attached to the socket. An implant was then placed.

Preoperative and Postoperative (5 months later) intraoral scans were superimposed with a digital software to assess the dimensional changes of the labial alveolar ridge. Linear changes at 1,3 and 5 mm from the gingival margin and mean linear changes in a specified Area Of Interest (AOI) were measured.

ELIGIBILITY:
Inclusion Criteria:

* medically healthy patients (ASA 1, ASA 2 categories) ,
* over 18 years old presenting with hopeless teeth due to extensive caries,
* cervical root fracture,
* vertical or oblique root fracture,
* multiple failed endodontic treatments,
* root resorption.

Exclusion Criteria:

* medically compromised patients (the ASA 3, ASA 4 and ASA5 categories)
* vertical root fracture involving the labial aspect of the root that will be retained,
* horizontal fracture of the root that is too far apically located
* presence of acute (active) periapical infection
* lack of sufficient bone to obtain implant primary stability apical and/or palatal to the extraction socket,
* ankylosed tooth which is positioned too apically in relation to the adjacent teeth,
* type 3 extraction sockets according to Elian and Tarnow extraction sockets classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-03 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
dimensional changes of the labial alveolar ridge in orofacial direction in millimeters using GOM Inspect software | 5 months
  Linear changes at 1,3 and 5 mm from the gingival margin and mean linear changes in a specified Area Of Interest (AOI) were measured.
Thickness of the labial plate of bone in millimeters on the preoperative CBCT radiograph | Preoperative
  On the preoperative CBCT scan, the thickness of the labial plate of bone was measured at the thickest part of its coronal third.The labial plate of bone was also checked for the presence of any radiographic coronal dehiscence and/or apical perforation by the root apex.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Nabawy, BDS, Principal Investigator — Alexandria university, Faculty of dentistry
Locations (1):
- Alexandria university, Faculty of dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be available at the end of the study
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: Requests to access IPD should be sent to the principal investigator by e-mail. All collected IPD will be sent to the other researchers by e-mail upon request.